CLINICAL TRIAL: NCT01355445
Title: International Randomized Phase II Trial of the Combination of Vincristine and Irinotecan With or Without Temozolomide (VI or VIT) in Children and Adults With Refractory or Relapsed Rhabdomyosarcoma
Brief Title: Vincristine and Irinotecan With or Without Temozolomide in Children and Adults With Refractory/Relapsed Rhabdomyosarcoma
Acronym: VIT-0910
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: SFCE (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIT-0910; 2010-023135-42 (EudraCT Number)
Record Dates: First submitted 2011-05-16; First posted 2011-05-18 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: RHABDOMYOSARCOMA
MeSH Terms: conditions — Rhabdomyosarcoma | interventions — Vincristine; Irinotecan; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vincristine / Irinotecan (Active Comparator): Vincristine, Irinotecan Vincristine :1.5 mg/m² (max 2mg), IV Irinotecan : Irinotecan 50 mg/m²/d, IV
  Interventions: Drug: Vincristine, Irinotecan
- Vincristine / Irinotecan / Temozolomide (Experimental): Vincristine, Irinotecan, Temozolomide
  Interventions: Drug: Vincristine, Irinotecan, Temozolomide

INTERVENTIONS:
Drug: Vincristine, Irinotecan — * D1 and D8: Vincristine 1.5 mg/m² (max 2mg) direct IV infusion (0.05 mg/kg for patient ≤ 10 kg)
  * D1 to D5: Irinotecan 50 mg/m²/d, IV
    1. cycle / 21 days
  Other Names: Vincristine-Irinotecan
  Arms: Vincristine / Irinotecan
Drug: Vincristine, Irinotecan, Temozolomide — * D1 to D5: Temozolomide 125 mg/m²/d, PO (the dose will be escalated to 150 mg/m²/day at cycle 2 for patients who do not experience > grade 3 toxicity of any kind)
  * D1 and D8: Vincristine 1.5 mg/m² (maximum 2mg) direct IV infusion (0.05 mg/kg for patient ≤ 10 kg)
  * D1 to D5: Irinotecan 50 mg/m²/d, IV
    1. cycle / 21 days
  Other Names: Vincristine-Irinotecan-Temozolomide
  Arms: Vincristine / Irinotecan / Temozolomide

SUMMARY:
This is an international open-label, randomized, multicenter phase II study of VIT and VI for the treatment of patients with recurrent or refractory rhabdomyosarcoma. The study will evaluate the safety and efficacy of these combinations in patients with recurrent or refractory rhabdomyosarcoma.

DETAILED DESCRIPTION:
The dose of vincristine will be 1.5 mg/m² or 0.05 mg/kg for patient ≤ 10 kg (maximum 2 mg) and will be administered by direct intravenous infusion on day 1 and 8 of each course, before irinotecan.

The dose of irinotecan will be 50 mg/m²/d. Irinotecan will be given intravenously over 1 hour on days 1-5 of each course, one hour following the administration of temozolomide.

In the absence of any contraindication (ie known allergies), treatment with oral cefixime 8 mg/kg once daily (maximum daily dose 400 mg) is recommended and will be started 2 days before chemotherapy until day 7.

Temozolomide will be given according to the randomization. The starting dose of temozolomide will be 125 mg/m²/d. The dose of temozolomide will be escalated to 150 mg/m²/day at cycle 2 for patients who do not experience > grade 3 toxicity of any kind. Temozolomide will be given orally, on an empty stomach, on days 1 through 5 of each course.

Dose reductions and/or administration delays will be performed using specific predefined rules to accommodate individual patient tolerance of treatment and to maintain optimal dose intensity.

ELIGIBILITY:
Inclusion Criteria:

* TUMOR CHARACTERISTICS :

  * Histologically or cytologically confirmed diagnosis of rhabdomyosarcoma (RMS) (new biopsy recommended)
  * Relapsed or refractory disease which has failed standard treatment approaches
  * Patients must have measurable disease defined as lesions that can be measured in 3 dimensions by medical imaging techniques such as CT or MRI. Ascites, pleural fluid, bone marrow disease and lesions seen on Tc scintigraphy or PET scan only are not considered measurable for these patients
* PATIENT CHARACTERISTICS :

  * Age > 6 months and ≤ 50 years
  * Karnofsky performance status (PS) 70-100% (for patients > 12 years of age) OR Lansky Play Score 70-100% (for patients ≤ 12 years of age)
  * Life expectancy ≥ 12 weeks
  * Adequate bone marrow function :

    * Absolute neutrophil count ≥ 1000/mm3; and ≥ 500/mm3 in case of bone marrow disease
    * Platelet count ≥ 100000/mm3 ; and ≥ 75000/mm3 in case of bone marrow disease (transfusion independent)
    * Hemoglobin ≥ 8.5 g/dl (transfusion allowed)
  * Adequate renal function

    * Serum creatinine ≤ 1.5 X ULN for age
    * If serum creatinine > 1.5 ULN, creatinine clearance (or radioisotope GFR) must be >70 ml/min/1.73 m²
  * Adequate hepatic function :

    * Total bilirubin ≤ 1.5 times upper limit of normal (ULN) for age, except if the patient is known to have Gilbert's syndrome
    * ALT and AST ≤ 2.5 times ULN for age
  * Negative pregnancy test in females with childbearing potential
  * Fertile patients must use effective contraception
  * No active > grade 2 diarrhea or uncontrolled infection
  * No other malignancy, including secondary malignancy
  * Patient affiliated with a health insurance system. Applicable for French patients only Written informed consent of patient and/or parents/guardians
* PRIOR or CONCURRENT THERAPY :

  * More than 3 weeks since prior radiation therapy to the site of any progressive lesion that will be identified as a target lesion to measure tumor response
  * At least 3 weeks since prior myelosuppressive therapy (6 weeks for nitrosourea. 2 weeks for vincristine, vinblastine, vinorelbine or low dose cyclophosphamide)
  * No concurrent enzyme-inducing anticonvulsants (EIAC), including phenytoin, phenobarbital or carbamazepine
  * No concurrent administration of any of the following: rifampicin, voriconazole,itraconazole, ketoconazole, aprepitant, St John's Wort
  * No prior irinotecan or temozolomide administration
  * Prior vincristine administration allowed
  * Concurrent palliative radiation therapy to sites allowed other than the main measurable target
  * Prior allo- or autologous SCT allowed

Exclusion Criteria:

* Inclusion criteria failure
* Concomitant anti-cancer treatment
* Know hypersensitivity to any component of study drugs or ingredients
* Pregnancy or breast feeding
* Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
* Neuromuscular disorders (e.g. Charcot-Marie Tooth disease)
* Uncontrolled intercurrent illness or active infection
* Unavailable for medical follow-up (geographic, social or psychological reasons)

Ages: 6 Months to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Objective tumour response and progression in each treatment arm. | at least 6 weeks (two cycles of treatment)
  The primary efficacy endpoint is defined as the proportion of patients who had a documented complete or partial tumour response occurring after the first 2 cycles of treatment which must be confirmed by a follow-up objective tumour assessment obtained within 4-5 weeks after the initial documentation.

SECONDARY OUTCOMES:
To assess the duration of tumor response in each treatment arm | During all the study
  The duration of tumour response is defined as the time from first documentation of objective tumour response to the first objective or clinical documentation of progression
To determine the time to tumor progression in each treatment arm | During all the study
  The time to tumor progression: the time from the date of first treatment administration to the date of first objective or clinical documentation of tumour progression or death due to any cause
To assess the time to treatment failure in each treatment arm | Before 1 year
  The time to treatment failure is defined as the time from the date of first treatment administration to the first documentation of tumour progression, discontinuation of study treatment before one year, or death, whichever occurs first
To assess the overall survival in each treament arm | During all the study
  The overall survival is defined as the time from the date of first treatment administration to date of death
To assess the safety profile and tolerability in each treatment arm | During all the study
  Safety parameters include adverse events and haematology and blood chemistry assays.
  Safety evaluations will include characterization of the frequency and severity of adverse events, complete blood cell counts with differential, serum chemistries and electrolytes, and change in weight and body surface area (BSA).

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie DEFACHELLES, MD, Principal Investigator — Centre Ocsar Lambret, Lille, France; Julia CHISHOLM, MD, Principal Investigator — Royal Marsden NHS Foundation Trust, Surrey, Uinted Kingdom; J.H.M. MD MERKS, Principal Investigator — Emma Children's Hospital, Amsterdam, The Netherlands; Michela CASANOVA, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale Tumori, Milano, Italy; Soledad GALLEGO, MDn, Principal Investigator — Hospital Materno - Infantil Vall D' Hebron, Barcelona, Spain
Locations (16):
- France (16):
  - CHU d'Amiens Picardie Site Sud, Amiens
  - Hôpital des Enfants, Groupe Hospitalier Pellegrin, Bordeaux
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - CHU, Hôpital d'Enfants de la Timone, Marseille
  - Hôpital Arnaud de Villeneuve - CHU, Montpellier
  - CHU, Hôpital Mère enfants, Nantes
  - Hôpital Armand Trousseau, Paris
  - Institut Curie, Paris
  - Hôpital Jean Bernard, Poitiers
  - CHU Rennes - Hôpital Sud, Rennes
  - CHU St Etienne - Hôpital Nord, Saint-Etienne
  - Hôpital des enfants, Toulouse
  - CHRU, Tours
  - CHRU Hôpital d'Enfants, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Defachelles AS, Bogart E, Casanova M, Merks JHM, Bisogno G, Calareso G, Gallego Melcon S, Gatz SA, Le Deley MC, McHugh K, Probst A, Rocourt N, van Rijn RR, Wheatley K, Minard-Colin V, Chisholm JC. Randomized Phase II Trial of Vincristine-Irinotecan With or Without Temozolomide, in Children and Adults With Relapsed or Refractory Rhabdomyosarcoma: A European Paediatric Soft Tissue Sarcoma Study Group and Innovative Therapies for Children With Cancer Trial. J Clin Oncol. 2021 Sep 20;39(27):2979-2990. doi: 10.1200/JCO.21.00124. Epub 2021 Aug 3. PMID 34343032